CLINICAL TRIAL: NCT01077674
Title: Comparison of Bispectral Index and Entropy With Electroencephalogram During Sevoflurane Anaesthesia
Brief Title: Comparison of Two Electroencephalogram (EEG)-Derived Indices With Electroencephalogram Signals
Status: Completed | Type: Observational
Sponsor: Arvi Yli-Hankala (Other)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Sponsor-Investigator, Arvi Yli-Hankala, Professor, Tampere University Hospital
Organization: Tampere University Hospital (Other)
Other Study IDs: Kotoe_03
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Anaesthesia; Surgery
Keywords: Electroencephalogram; Entropy; BIS; Sevoflurane

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Entropy - BIS: Patients undergoing surgery in sevoflurane anaesthesia.

SUMMARY:
Bispectral Index (BIS) and Entropy indices will be compared with each other, and to raw EEG signals in patients receiving sevoflurane anaesthesia. BIS and Entropy numbers often differ significantly from each other during surgery, and the reason for this has not been studied in detail, therefore remaining only poorly understood. BIS and Entropy, together with multi-channel EEG, will be collected and analyzed later on. Course of anaesthesia and surgery will be annotated. All relevant information from anaesthesia monitor will be collected on computer.

ELIGIBILITY:
Inclusion Criteria:

* Planned surgery necessitating general anaesthesia
* Expected duration of anaesthesia 30 min or more
* Need of endotracheal intubation
* ASA status 1, 2 or 3

Exclusion Criteria:

* Significant disorders of the autonomic or central nervous system
* Family history of malignant hyperthermia
* Clinical history of anaphylactic reaction against inhaled anaesthetics
* Disability to communicate with Finnish language

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Middle aged and elderly surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Morphology of electroencephalogram during discrepancy between Entropy and BIS index values | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Arvi Yli-Hankala, MD, Study Chair — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Derived] Aho AJ, Kamata K, Jantti V, Kulkas A, Hagihira S, Huhtala H, Yli-Hankala A. Comparison of Bispectral Index and Entropy values with electroencephalogram during surgical anaesthesia with sevoflurane. Br J Anaesth. 2015 Aug;115(2):258-66. doi: 10.1093/bja/aev206. Epub 2015 Jul 1. PMID 26137969